CLINICAL TRIAL: NCT03442088
Title: An Investigator Initiated Study of Monocyte Biomarkers in Moderate to Severe Plaque Psoriasis Subjects Treated With Apremilast
Brief Title: Monocyte Biomarkers in Moderate to Severe Plaque Psoriasis Subjects Treated With Apremilast
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-17-33
Record Dates: First submitted 2017-10-11; First posted 2018-02-22 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Intervention Model Description: This is an open label pilot study of the impact of treatment with standard dosing of APM for 16 weeks on AM-endotype psoriasis patients, identified by elevated (>150% of normal): 1.) Intermediate (CD14++CD16+) monocytes % of cells in circulation, or 2.) circulating monocyte doublets % of adherent monocyte-monocyte pairs, or 3.) circulating monocyte-platelet aggregates (MPA) % monocytes adherent to platelets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Apremilast for Treatment of Psoriasis with the AM-endotype (Experimental): Psoriasis patients with the AM-endotype will be followed during treatment over 16 weeks with 5 monthly individual blood draws will be enrolled.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast will be given as approved by the FDA for the treatment of moderate to severe plaque psoriasis. An initial dosage titration from Day 1 (10mg) to Day 5 (30mg). Following the titration, the recommended maintenance dosage of 30 mg twice daily taken orally starting on Day 6 will be dispensed, as per labeled indication.
  Other Names: Otezla

SUMMARY:
This is an open label pilot study of the impact of treatment with standard dosing of Otezla for 16 weeks on AM-endotype psoriasis patients, identified by elevated (>150% of normal): 1.) Intermediate (CD14++CD16+) monocytes, or 2.) circulating monocyte doublets, or 3.) circulating monocyte-platelet aggregates (MPA).

Approximately 25 psoriasis patients with the AM-endotype will be followed during treatment over 16 weeks with 4 monthly individual blood draws will be enrolled. All treated psoriasis subjects will receive apremilast through Week 16.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ≥ 18 and < 60 years of age at the time of signing the informed consent document.
2. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Patients must exhibit AM-endotype psoriasis patients, identified by elevated (>150% of normal) levels of any one of the following criteria: 1.) Intermediate (CD14++CD16+) monocytes, or 2.) circulating monocyte doublets, or 3.) circulating monocyte-platelet aggregates (MPA).
5. Diagnosis of chronic plaque psoriasis for at least 12 months prior to Screening.
6. Have moderate to severe plaque psoriasis at Screening and Baseline as defined by a. BSA ≥5% b. sPGA ≥3 (moderate to severe)
7. Must be a candidate for phototherapy and systemic (including Otezla) therapy.
8. Must be in good health (except for psoriasis) as judged by the Investigator, based on medical history and physical examination.
9. Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy;

OR

Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on investigational product and for at least 28 days after the last dose of investigational product.

Exclusion Criteria:

* 1. Other than psoriasis, history of any clinically significant (as determined by the Investigator) cardiac (clinically advanced cardiovascular disease including; Stent, past history of MI, thrombotic event or arterial calcification), endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major uncontrolled disease.

  2. Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.

  3. Any condition, including other inflammatory diseases or dermatologic conditions that confound the ability to interpret data from the study.

  4. Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.

  5. Pregnant or breast feeding.

  6. Have failed more than 3 systemic agents for treatment of psoriasis.

  7. History of allergy to any component of Apremilast.

  8. Hepatitis B surface antigen positive at Screening.

  9. Anti-hepatitis C antibody positive at Screening.

  10. Had a serious infection (including, but not limited to, hepatitis, pneumonia, sepsis, cellulitis, meningitis or pyelonephritis) or have been hospitalized for an infection. Subject must be cured of infection > 4 weeks before Screening.

  11. Have a history of, or ongoing, chronic or recurrent infectious disease, including, but not limited to, chronic renal infection, chronic chest infection (e.g., bronchiectasis), sinusitis, recurrent urinary tract infection (e.g., recurrent pyelonephritis, chronic nonremitting cystitis), an open, draining, or infected skin wound or ulcer.

  12. Had a Bacillus Calmette-Guérin (BCG) vaccination within 1 year prior to screening.

  13. History of positive human immunodeficiency virus (HIV), or have congenital or acquired immunodeficiency (e.g., common variable immunodeficiency disease).

  14. Active substance abuse or a history of substance abuse within 6 months prior to Screening.

  15. Bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of Screening. Any treatment and cure for such infections must have been completed at least 4 weeks prior to Screening.

  16. Malignancy or history of malignancy, except for:
  1. treated [i.e., cured] basal cell or squamous cell in situ skin carcinomas;
  2. treated [i.e., cured] cervical intraepithelial neoplasia [CIN] or carcinoma in situ of the cervix with no evidence of recurrence within the previous 5 years.

     17. Topical therapy within 2 weeks of study entry (including, but not limited to, topical corticosteroids, retinoids or vitamin D analog preparations, tacrolimus, pimecrolimus, or anthralin/dithranol). Exceptions: low-potency corticosteroids to cyclosporine, corticosteroids, methotrexate, retinoids, mycophenolate, thioguanine, hydroxyurea, sirolimus, sulfasalazine, azathioprine, fumaric acid esters) will be allowed as background therapy and restricted to treatment of the face, axillae, and groin in accordance with the manufacturers' suggested usage during the course of the study (this restricted usage should be documented). Subjects with scalp psoriasis will be permitted to use coal tar shampoo and/or salicylic acid scalp preparations on scalp lesions. An unmedicated skin moisturizer (eg, Eucerin®) will be also permitted for body lesions only. Subjects should not use these topical treatments within 24 hours prior to the clinic visit.

     18. Systemic therapy for psoriasis within 4 weeks prior to study entry (including, but not limited to, cyclosporine, corticosteroids, methotrexate, retinoids, mycophenolate, thioguanine, hydroxyurea, sirolimus, sulfasalazine, azathioprine, and fumaric acid esters).

     19. Use of phototherapy within 4 weeks prior to study entry.

     20. Use of any investigational drug within 4 weeks prior to study entry, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).

     21. Prolonged sun exposure or use of tanning booths or other ultraviolet (UV) light sources.

     22. Prior treatment with Apremilast

     23. Inability to wash out from any topical treatment(s) (two weeks prior to entering the study) or all systemic therapies, including orals and biologics (e.g., TNF inhibitors IL-17 inhibitors, IL-12/23 inhibitors, 4 weeks).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Cooper, MD, Study Chair — University Hospitals Cleveland Medical Center; Neil Korman, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ackermann C, Kavanaugh A. Economic burden of psoriatic arthritis. Pharmacoeconomics. 2008;26(2):121-9. doi: 10.2165/00019053-200826020-00003. PMID 18198932
- [Background] Feldman SR, Evans C, Russell MW. Systemic treatment for moderate to severe psoriasis: estimates of failure rates and direct medical costs in a north-eastern US managed care plan. J Dermatolog Treat. 2005 Feb;16(1):37-42. doi: 10.1080/09546630510025941. PMID 15897166
- [Background] Fowler JF, Duh MS, Rovba L, Buteau S, Pinheiro L, Lobo F, Sung J, Doyle JJ, Swensen A, Mallett DA, Kosicki G. The impact of psoriasis on health care costs and patient work loss. J Am Acad Dermatol. 2008 Nov;59(5):772-80. doi: 10.1016/j.jaad.2008.06.043. PMID 19119095
- [Background] Hazard E, Cherry SB, Lalla D, Woolley JM, Wilfehrt H, Chiou CF. Clinical and economic burden of psoriasis. Manag Care Interface. 2006 Apr;19(4):20-6. PMID 16689023
- [Background] Kimball AB, Guerin A, Tsaneva M, Yu AP, Wu EQ, Gupta SR, Bao Y, Mulani PM. Economic burden of comorbidities in patients with psoriasis is substantial. J Eur Acad Dermatol Venereol. 2011 Feb;25(2):157-63. doi: 10.1111/j.1468-3083.2010.03730.x. Epub 2010 Jun 17. PMID 20561129
- [Background] Davidovici BB, Sattar N, Prinz J, Puig L, Emery P, Barker JN, van de Kerkhof P, Stahle M, Nestle FO, Girolomoni G, Krueger JG. Psoriasis and systemic inflammatory diseases: potential mechanistic links between skin disease and co-morbid conditions. J Invest Dermatol. 2010 Jul;130(7):1785-96. doi: 10.1038/jid.2010.103. Epub 2010 May 6. PMID 20445552
- [Background] Kim N, Thrash B, Menter A. Comorbidities in psoriasis patients. Semin Cutan Med Surg. 2010 Mar;29(1):10-5. doi: 10.1016/j.sder.2010.01.002. PMID 20430302
- [Background] Gelfand JM, Shin DB, Neimann AL, Wang X, Margolis DJ, Troxel AB. The risk of lymphoma in patients with psoriasis. J Invest Dermatol. 2006 Oct;126(10):2194-201. doi: 10.1038/sj.jid.5700410. Epub 2006 Jun 1. PMID 16741509
- [Background] Mehta NN, Azfar RS, Shin DB, Neimann AL, Troxel AB, Gelfand JM. Patients with severe psoriasis are at increased risk of cardiovascular mortality: cohort study using the General Practice Research Database. Eur Heart J. 2010 Apr;31(8):1000-6. doi: 10.1093/eurheartj/ehp567. Epub 2009 Dec 27. PMID 20037179
- [Background] Kimball AB, Jacobson C, Weiss S, Vreeland MG, Wu Y. The psychosocial burden of psoriasis. Am J Clin Dermatol. 2005;6(6):383-92. doi: 10.2165/00128071-200506060-00005. PMID 16343026
- [Background] Au L, Meisch JP, Das LM, Binko AM, Boxer RS, Wen AM, Steinmetz NF, Lu KQ. Suppression of Hyperactive Immune Responses Protects against Nitrogen Mustard Injury. J Invest Dermatol. 2015 Dec;135(12):2971-2981. doi: 10.1038/jid.2015.322. Epub 2015 Aug 19. PMID 26288355
- [Background] Ziegler-Heitbrock HW. Heterogeneity of human blood monocytes: the CD14+ CD16+ subpopulation. Immunol Today. 1996 Sep;17(9):424-8. doi: 10.1016/0167-5699(96)10029-3. No abstract available. PMID 8854561
- [Background] Martinez FO. The transcriptome of human monocyte subsets begins to emerge. J Biol. 2009;8(11):99. doi: 10.1186/jbiol206. Epub 2009 Dec 23. PMID 20067595
- [Background] Ancuta P, Liu KY, Misra V, Wacleche VS, Gosselin A, Zhou X, Gabuzda D. Transcriptional profiling reveals developmental relationship and distinct biological functions of CD16+ and CD16- monocyte subsets. BMC Genomics. 2009 Aug 27;10:403. doi: 10.1186/1471-2164-10-403. PMID 19712453
- [Background] Wong KL, Tai JJ, Wong WC, Han H, Sem X, Yeap WH, Kourilsky P, Wong SC. Gene expression profiling reveals the defining features of the classical, intermediate, and nonclassical human monocyte subsets. Blood. 2011 Aug 4;118(5):e16-31. doi: 10.1182/blood-2010-12-326355. Epub 2011 Jun 7. PMID 21653326
- [Background] Zawada AM, Rogacev KS, Rotter B, Winter P, Marell RR, Fliser D, Heine GH. SuperSAGE evidence for CD14++CD16+ monocytes as a third monocyte subset. Blood. 2011 Sep 22;118(12):e50-61. doi: 10.1182/blood-2011-01-326827. Epub 2011 Jul 29. PMID 21803849
- [Background] Zawada AM, Rogacev KS, Schirmer SH, Sester M, Bohm M, Fliser D, Heine GH. Monocyte heterogeneity in human cardiovascular disease. Immunobiology. 2012 Dec;217(12):1273-84. doi: 10.1016/j.imbio.2012.07.001. Epub 2012 Jul 25. PMID 22898391
- [Background] Ziegler-Heitbrock L, Ancuta P, Crowe S, Dalod M, Grau V, Hart DN, Leenen PJ, Liu YJ, MacPherson G, Randolph GJ, Scherberich J, Schmitz J, Shortman K, Sozzani S, Strobl H, Zembala M, Austyn JM, Lutz MB. Nomenclature of monocytes and dendritic cells in blood. Blood. 2010 Oct 21;116(16):e74-80. doi: 10.1182/blood-2010-02-258558. Epub 2010 Jul 13. PMID 20628149
- [Background] Geissmann F, Jung S, Littman DR. Blood monocytes consist of two principal subsets with distinct migratory properties. Immunity. 2003 Jul;19(1):71-82. doi: 10.1016/s1074-7613(03)00174-2. PMID 12871640
- [Background] Auffray C, Sieweke MH, Geissmann F. Blood monocytes: development, heterogeneity, and relationship with dendritic cells. Annu Rev Immunol. 2009;27:669-92. doi: 10.1146/annurev.immunol.021908.132557. PMID 19132917
- [Background] Shantsila E, Wrigley B, Tapp L, Apostolakis S, Montoro-Garcia S, Drayson MT, Lip GY. Immunophenotypic characterization of human monocyte subsets: possible implications for cardiovascular disease pathophysiology. J Thromb Haemost. 2011 May;9(5):1056-66. doi: 10.1111/j.1538-7836.2011.04244.x. PMID 21342432
- [Background] Gallego C, Golenbock D, Gomez MA, Saravia NG. Toll-like receptors participate in macrophage activation and intracellular control of Leishmania (Viannia) panamensis. Infect Immun. 2011 Jul;79(7):2871-9. doi: 10.1128/IAI.01388-10. Epub 2011 Apr 25. PMID 21518783
- [Background] Cao LY, Soler DC, Debanne SM, Grozdev I, Rodriguez ME, Feig RL, Carman TL, Gilkeson RC, Orringer CE, Kern EF, McCormick TS, Cooper KD, Korman NJ. Psoriasis and cardiovascular risk factors: increased serum myeloperoxidase and corresponding immunocellular overexpression by Cd11b(+) CD68(+) macrophages in skin lesions. Am J Transl Res. 2013 Dec 1;6(1):16-27. eCollection 2013. PMID 24349618
- [Background] Tapp LD, Shantsila E, Wrigley BJ, Pamukcu B, Lip GY. The CD14++CD16+ monocyte subset and monocyte-platelet interactions in patients with ST-elevation myocardial infarction. J Thromb Haemost. 2012 Jul;10(7):1231-41. doi: 10.1111/j.1538-7836.2011.04603.x. PMID 22212813
- [Background] Tapp LD, Shantsila E, Wrigley BJ, Montoro-Garcia S, Lip GY. TLR4 expression on monocyte subsets in myocardial infarction. J Intern Med. 2013 Mar;273(3):294-305. doi: 10.1111/joim.12011. Epub 2012 Dec 28. PMID 23121518
- [Background] Garcia-Rodriguez S, Arias-Santiago S, Perandres-Lopez R, Castellote L, Zumaquero E, Navarro P, Buendia-Eisman A, Ruiz JC, Orgaz-Molina J, Sancho J, M Zubiaur. Increased gene expression of Toll-like receptor 4 on peripheral blood mononuclear cells in patients with psoriasis. J Eur Acad Dermatol Venereol. 2013 Feb;27(2):242-50. doi: 10.1111/j.1468-3083.2011.04372.x. PMID 23457721
- [Background] Benoit S, Toksoy A, Ahlmann M, Schmidt M, Sunderkotter C, Foell D, Pasparakis M, Roth J, Goebeler M. Elevated serum levels of calcium-binding S100 proteins A8 and A9 reflect disease activity and abnormal differentiation of keratinocytes in psoriasis. Br J Dermatol. 2006 Jul;155(1):62-6. doi: 10.1111/j.1365-2133.2006.07198.x. PMID 16792753
- [Background] Funderburg NT, Zidar DA, Shive C, Lioi A, Mudd J, Musselwhite LW, Simon DI, Costa MA, Rodriguez B, Sieg SF, Lederman MM. Shared monocyte subset phenotypes in HIV-1 infection and in uninfected subjects with acute coronary syndrome. Blood. 2012 Nov 29;120(23):4599-608. doi: 10.1182/blood-2012-05-433946. Epub 2012 Oct 11. PMID 23065151
- [Background] Chiu YG, Shao T, Feng C, Mensah KA, Thullen M, Schwarz EM, Ritchlin CT. CD16 (FcRgammaIII) as a potential marker of osteoclast precursors in psoriatic arthritis. Arthritis Res Ther. 2010;12(1):R14. doi: 10.1186/ar2915. Epub 2010 Jan 26. PMID 20102624
- [Background] Moniuszko M, Bodzenta-Lukaszyk A, Kowal K, Lenczewska D, Dabrowska M. Enhanced frequencies of CD14++CD16+, but not CD14+CD16+, peripheral blood monocytes in severe asthmatic patients. Clin Immunol. 2009 Mar;130(3):338-46. doi: 10.1016/j.clim.2008.09.011. Epub 2008 Oct 25. PMID 18952503
- [Background] Mysliwska J, Smardzewski M, Marek-Trzonkowska N, Mysliwiec M, Raczynska K. Expansion of CD14+CD16+ monocytes producing TNF-alpha in complication-free diabetes type 1 juvenile onset patients. Cytokine. 2012 Oct;60(1):309-17. doi: 10.1016/j.cyto.2012.03.010. Epub 2012 Apr 7. PMID 22484242
- [Background] Hanai H, Iida T, Takeuchi K, Watanabe F, Yamada M, Kikuyama M, Maruyama Y, Iwaoka Y, Hirayama K, Nagata S, Takai K. Adsorptive depletion of elevated proinflammatory CD14+CD16+DR++ monocytes in patients with inflammatory bowel disease. Am J Gastroenterol. 2008 May;103(5):1210-6. doi: 10.1111/j.1572-0241.2007.01714.x. Epub 2008 Jan 2. PMID 18177452
- [Background] Skrzeczynska J, Kobylarz K, Hartwich Z, Zembala M, Pryjma J. CD14+CD16+ monocytes in the course of sepsis in neonates and small children: monitoring and functional studies. Scand J Immunol. 2002 Jun;55(6):629-38. doi: 10.1046/j.1365-3083.2002.01092.x. PMID 12028567
- [Background] Blumenstein M, Boekstegers P, Fraunberger P, Andreesen R, Ziegler-Heitbrock HW, Fingerle-Rowson G. Cytokine production precedes the expansion of CD14+CD16+ monocytes in human sepsis: a case report of a patient with self-induced septicemia. Shock. 1997 Jul;8(1):73-5. doi: 10.1097/00024382-199707000-00012. PMID 9249916
- [Background] Fingerle G, Pforte A, Passlick B, Blumenstein M, Strobel M, Ziegler-Heitbrock HW. The novel subset of CD14+/CD16+ blood monocytes is expanded in sepsis patients. Blood. 1993 Nov 15;82(10):3170-6. PMID 7693040
- [Background] Schlitt A, Heine GH, Blankenberg S, Espinola-Klein C, Dopheide JF, Bickel C, Lackner KJ, Iz M, Meyer J, Darius H, Rupprecht HJ. CD14+CD16+ monocytes in coronary artery disease and their relationship to serum TNF-alpha levels. Thromb Haemost. 2004 Aug;92(2):419-24. doi: 10.1160/TH04-02-0095. PMID 15269840
- [Background] Rogacev KS, Cremers B, Zawada AM, Seiler S, Binder N, Ege P, Grosse-Dunker G, Heisel I, Hornof F, Jeken J, Rebling NM, Ulrich C, Scheller B, Bohm M, Fliser D, Heine GH. CD14++CD16+ monocytes independently predict cardiovascular events: a cohort study of 951 patients referred for elective coronary angiography. J Am Coll Cardiol. 2012 Oct 16;60(16):1512-20. doi: 10.1016/j.jacc.2012.07.019. Epub 2012 Sep 19. PMID 22999728
- [Background] Wrigley BJ, Shantsila E, Tapp LD, Lip GY. CD14++CD16+ monocytes in patients with acute ischaemic heart failure. Eur J Clin Invest. 2013 Feb;43(2):121-30. doi: 10.1111/eci.12023. Epub 2012 Dec 14. PMID 23240665
- [Background] Brunner PM, Koszik F, Reininger B, Kalb ML, Bauer W, Stingl G. Infliximab induces downregulation of the IL-12/IL-23 axis in 6-sulfo-LacNac (slan)+ dendritic cells and macrophages. J Allergy Clin Immunol. 2013 Nov;132(5):1184-1193.e8. doi: 10.1016/j.jaci.2013.05.036. Epub 2013 Jul 26. PMID 23890755
- [Background] Golden JB, Groft SG, Squeri MV, Debanne SM, Ward NL, McCormick TS, Cooper KD. Chronic Psoriatic Skin Inflammation Leads to Increased Monocyte Adhesion and Aggregation. J Immunol. 2015 Sep 1;195(5):2006-18. doi: 10.4049/jimmunol.1402307. Epub 2015 Jul 29. PMID 26223654
- [Background] Schafer PH, Parton A, Gandhi AK, Capone L, Adams M, Wu L, Bartlett JB, Loveland MA, Gilhar A, Cheung YF, Baillie GS, Houslay MD, Man HW, Muller GW, Stirling DI. Apremilast, a cAMP phosphodiesterase-4 inhibitor, demonstrates anti-inflammatory activity in vitro and in a model of psoriasis. Br J Pharmacol. 2010 Feb;159(4):842-55. doi: 10.1111/j.1476-5381.2009.00559.x. Epub 2009 Dec 24. PMID 20050849
- [Background] Singri P, West DP, Gordon KB. Biologic therapy for psoriasis: the new therapeutic frontier. Arch Dermatol. 2002 May;138(5):657-63. doi: 10.1001/archderm.138.5.657. PMID 12020229
- [Background] Chaudhari U, Romano P, Mulcahy LD, Dooley LT, Baker DG, Gottlieb AB. Efficacy and safety of infliximab monotherapy for plaque-type psoriasis: a randomised trial. Lancet. 2001 Jun 9;357(9271):1842-7. doi: 10.1016/s0140-6736(00)04954-0. PMID 11410193
- [Background] Krueger GG, Langley RG, Leonardi C, Yeilding N, Guzzo C, Wang Y, Dooley LT, Lebwohl M; CNTO 1275 Psoriasis Study Group. A human interleukin-12/23 monoclonal antibody for the treatment of psoriasis. N Engl J Med. 2007 Feb 8;356(6):580-92. doi: 10.1056/NEJMoa062382. PMID 17287478
- [Background] Desai SB, Furst DE. Problems encountered during anti-tumour necrosis factor therapy. Best Pract Res Clin Rheumatol. 2006 Aug;20(4):757-90. doi: 10.1016/j.berh.2006.06.002. PMID 16979537

RESULTS

PARTICIPANT FLOW:
Groups:
- Apremilast for Treatment of Psoriasis With the AM-endotype: Psoriasis patients with the AM-endotype will be followed during treatment over 16 weeks with 5 monthly individual blood draws will be enrolled.
  Apremilast: Apremilast will be given as approved by the FDA for the treatment of moderate to severe plaque psoriasis. An initial dose titration from Day 1 (10mg) to Day 5 (30mg). Following titration, the recommended maintenance dosage of 30 mg twice daily taken orally starting on Day 6 will be dispensed, as per labeled indication.
Period: Overall Study
Arm/Group | Apremilast for Treatment of Psoriasis With the AM-endotype
Started | 28
Completed | 23
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Apremilast for Treatment of Psoriasis With the AM-endotype
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 22
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Will be to Evaluate Change in Aberrant Inflammatory Profiles of Activated Blood Monocytes (Aberrant-monocyte Endotype Patients (AM-endotype).
Description: For each subject, we will identify a target biomarker of abnormally elevated monocytes, among 1.) intermediate, or 2.) doublets, or 3.) platelet doubles. Each subject will thus have one identified monocyte biomarker for which relative percent change will be its basis for analysis in the primary outcome measure. We will specifically assess change from baseline to 16 weeks by computing relative percent reduction for each subject being treated. Note for example that a change of 1.5% to 1.2% is (1 - (1.2/1.5))*100% = 20% reduction. The median and other summary statistics of these percent change values will be computed. Wilcoxon's signed rank test will be used to evaluate the null hypothesis of the median percent change being 0.
Time Frame: Baseline, Week 16
Population: 1 subject missed interim visits, so data was not analyzed for this one participant.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Apremilast for Treatment of Psoriasis With the AM-endotype
Number analyzed (Participants) | 22
Percent change
  Baseline | 0.5665 (0.5135)
  Week 16 | 0.1715 (0.2635)
Statistical Analysis 1: Comparison: Apremilast for Treatment of Psoriasis With the AM-endotype; Test type: Other; p = 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.272

2. Secondary Outcome: Change in Serum Myeloperoxidase
Description: To assess change in serum myeloperoxidase in the identified patient AM-endotype computing relative percent reduction for each subject being treated and serum marker. The median and other summary statistics of these percent change values will be computed
Time Frame: Baseline, Week 16
Population: Analysis was only done on participants had complete data sets including sequencing.
Measure: Mean (Standard Deviation); unit: Pg/mL
Arm/Group | Apremilast for Treatment of Psoriasis With the AM-endotype
Number analyzed (Participants) | 17
Pg/mL
  Baseline | 24198 (3835)
  Week 16 | 24294 (4722)
Statistical Analysis 1: Comparison: Apremilast for Treatment of Psoriasis With the AM-endotype; Test type: Other; p = 0.934, t-test, 2 sided; Mean Difference (Final Values) = 95.98, 95% CI 2-sided [-2324 to 2516]

3. Secondary Outcome: Change in TNF Alpha
Description: To assess change in in the identified patient AM-endotype computing relative percent reduction for each subject being treated and serum marker. The median and other summary statistics of these percent change values will be computed
Time Frame: Baseline, Week 16
Population: Analysis was only done on participants had complete data sets including sequencing.
Measure: Mean (Standard Deviation); unit: Pg/mL
Arm/Group | Apremilast for Treatment of Psoriasis With the AM-endotype
Number analyzed (Participants) | 17
Pg/mL
  Baseline | 14.95 (4.017)
  Week 16 | 14.26 (3.383)
Statistical Analysis 1: Comparison: Apremilast for Treatment of Psoriasis With the AM-endotype; Test type: Other; p = 0.1632, t-test, 2 sided; Mean Difference (Final Values) = -0.6878, 95% CI 2-sided [-1.685 to 0.3097]

4. Secondary Outcome: Change in IL-17
Description: To assess change in IL-17 in the identified patient AM-endotype computing relative percent reduction for each subject being treated and serum marker. The median and other summary statistics of these percent change values will be computed
Time Frame: Baseline, Week 16
Population: Analysis was only done on participants had complete data sets including sequencing.
Measure: Mean (Standard Deviation); unit: Pg/mL
Arm/Group | Apremilast for Treatment of Psoriasis With the AM-endotype
Number analyzed (Participants) | 17
Pg/mL
  Baseline | 1.513 (5.76)
  Week 16 | -0.8315 (5.824)
Statistical Analysis 1: Comparison: Apremilast for Treatment of Psoriasis With the AM-endotype; Test type: Other; p = 0.1063, t-test, 2 sided; Mean Difference (Final Values) = -2.344, 95% CI 2-sided [-5.248 to 0.5992]

5. Secondary Outcome: Change in Tissue Factor
Description: To assess change in Tissue Factor in the identified patient AM-endotype computing relative percent reduction for each subject being treated and serum marker. The median and other summary statistics of these percent change values will be computed
Time Frame: Baseline, Week 16
Population: Analysis was only done on participants had complete data sets including sequencing.
Measure: Mean (Standard Deviation); unit: Pg/mL
Arm/Group | Apremilast for Treatment of Psoriasis With the AM-endotype
Number analyzed (Participants) | 17
Pg/mL
  Baseline | 72.28 (23.72)
  Week 16 | 75.52 (28.03)
Statistical Analysis 1: Comparison: Apremilast for Treatment of Psoriasis With the AM-endotype; Test type: Other; p = 0.5611, t-test, 2 sided; Mean Difference (Final Values) = 3.24, 95% CI 2-sided [-8.333 to 14.81]

6. Other Pre Specified Outcome: Evaluate Median Changes in Flow Cytometric Quantification of Monocytes
Description: To assess change in quantitation of additional monocyte and neutrophil markers, including CD18/CD11b and NETotic neutrophils by computing relative percent reduction in circulating CD18/CD11b and NETotic neutrophils for each subject being treated.
Time Frame: 16 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Monocyte Transcriptome Biomarkers
Description: To assess change in expression levels of monocyte transcriptome biomarkers using quantitative PCR to measure changes from baseline to 16 weeks in identified monocyte genes.
Time Frame: 16 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Percent Change in Dermatology Life Quality Index (DLQI)
Description: Calculate the percent change in Dermatology Life Quality Index (DLQI) from baseline to 16 weeks in patients.
Time Frame: 16 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Percent Change Between Work Productivity and Activity Impairment Questionnaire: Psoriasis (WPAI: PSO
Description: Calculate the percent change Work Productivity and Activity Impairment Questionnaire: Psoriasis (WPAI: PSO) from baseline to 16 weeks in patients treated with apremilast 30 mg BID
Time Frame: 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: While patients were on treatment, 16 weeks.
Arm/Group | Apremilast for Treatment of Psoriasis With the AM-endotype
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 13/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast for Treatment of Psoriasis With the AM-endotype (N=28)
Nausea (Gastrointestinal disorders) | 1 (5)
Diarrhea (Gastrointestinal disorders) | 1 (6)
Sinus/viral infection (Infections and infestations) | 1 (3)
Arthroscopic procedure (Surgical and medical procedures) | 1 (1)
Contact dermatitis to watch (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis flare (Skin and subcutaneous tissue disorders) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
COVID (Infections and infestations) | 1 (1)
Headache (General disorders) | 1 (2)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Sprained ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Itchiness (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT03442088/Prot_SAP_000.pdf